CLINICAL TRIAL: NCT03583684
Title: Neuroimaging Predictors of Improvement to Pivotal Response Treatment (PRT) in Young Children With Autism
Acronym: PRT-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-46131; 1R21DC016089-01A1 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-07-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Pivotal Response Treatment; Imaging
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pivotal Response Treatment Program (PRT-P) (Experimental): The Pivotal Response Treatment Program (PRT-P) will consist of 3 parent-only sessions (60-90 min) and 13 family sessions with the parent and child (60-90 min). These 16 sessions are once per week over a 16 week period.
  Interventions: Behavioral: Pivotal Response Treatment Program (PRT-P)
- Delayed Treatment Group (DTG) (No Intervention): Child continues stable treatments as usual in the community.

INTERVENTIONS:
Behavioral: Pivotal Response Treatment Program (PRT-P) — The Pivotal Response Treatment Program (PRT-P) will consist of 3 parent-only sessions (60-90 min) and 13 family sessions with the parent and child (60-90 min). These 16 sessions are once per week over a 16 week period.
  Other Names: Pivotal Response Treatment
  Arms: Pivotal Response Treatment Program (PRT-P)

SUMMARY:
Autism spectrum disorder (ASD) is a very heterogeneous disorder with limited empirically validated behavioral and biological interventions. The goal of this pilot investigation is to apply a biologically-based approach to identify predictors of treatment response in children with ASD who are receiving Pivotal Response Treatment (PRT), an evidence-based behavioral intervention. Specifically, the investigators propose to identify neuroimaging biomarkers of treatment response to a PRT program (PRT-P) targeting language deficits in young children with ASD who will be randomized to either PRT-P or to a delayed treatment group (DTG).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Spectrum Disorder (ASD) based on clinical interview and Diagnostic and Statistical Manual, 5th edition (DSM-5) and confirmed using the Autism Diagnostic Interview Revised (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS) and/or Brief Observation of Symptoms of Autism (BOSA) and/or Childhood Autism Rating Scale- Second Edition (CARS-2).
* Outpatients between 2.0 and 4.11 years of age of either gender,
* Children of all cognitive levels will be included as long as they are able to participate in the testing procedures to the extent that valid standard scores can be obtained
* Language delay as measured by the Preschool Language Scale, 5th Edition (PLS-5) [at least 1 standard deviation behind for children age 2 and 3 years; and 2 standard deviations behind for children age 4],
* Stable psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements with no anticipated changes during study participation,
* Stable treatment [Applied Behavior Analysis (ABA), Floortime, or other interventions], speech therapy, and school placement for at least 1 month prior to baseline measurements with no expected changes during study participation,
* No more than 60 minutes of 1:1 speech therapy per week,
* The child's exposure to the English language must be sufficient that administration of standardized tests in English is appropriate for measuring progress,
* The availability of at least one parent who can consistently participate in the training sessions and related activities, and
* Successful completion of baseline brain scan.

Exclusion Criteria:

* Current or life-time diagnosis of severe psychiatric disorder (e.g., bipolar disorder),
* Genetic abnormality (e.g., Fragile X)
* Presence of active medical problem (e.g., unstable seizure disorder),
* Receiving more than 15 hours of in home 1:1 Applied Behavior Analysis (ABA) per week
* Magnetic Resonance (MR) contraindication (e.g., the presence of ferrous metal), or
* Previous adequate Pivotal Response Treatment (PRT) trial.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Child Utterances During a Structured Lab Observation (SLO) | Baseline, 16 Weeks

SECONDARY OUTCOMES:
Change on MacArthur-Bates Communication Development Inventory (CDI) | Baseline, 16 Weeks

OTHER OUTCOMES:
Change on Preschool Language Scale, 5th Edition (PLS-5) | Baseline, 16 Weeks
Change on Mullen Scales of Early Learning | Baseline, 16 Weeks
Change on Vineland Adaptive Behaviors Scales, 3rd Edition | Baseline, 16 Weeks
Change on Clinical Global Impressions Scale (CGI) | Baseline, 16 Weeks
Change on the Brief Observation of Social Communication Change (BOSCC) direct child observation assessment | Baseline, 16 Weeks
Change on Parent Stress Index (PSI) | Baseline, 16 Weeks
Change on Family Empowerment Scale (FES) | Baseline, 16 Weeks
Change on General Self Efficacy Scale (GSES) | Baseline, 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified clinical data to the NIMH Data Archive (NDA) data repository.
URL: https://nda.nih.gov/contribute/sharing-regimen.html